CLINICAL TRIAL: NCT06670274
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled, First-in-Human Dose Escalation Study of HC002 to Evaluate Safety, Tolerability, and Pharmacokinetics in Healthy Adult Volunteers
Brief Title: A Dose Escalating Study of HC002 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Holoclara Aus Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC002-001-24
Record Dates: First submitted 2024-10-21; First posted 2024-11-01 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Disease; Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 SAD (Experimental)
  Interventions: Drug: HC002 SAD
- Part 2 MAD (Experimental)
  Interventions: Drug: HC002 MAD
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HC002 SAD — Part 1 will enroll 32 participants across 4 cohorts.
  Route of administration: Oral Dose interval and frequency: Single oral dose range across 4 cohorts.
  Arms: Part 1 SAD
Drug: HC002 MAD — Part 2 will enroll 24 participants across 3 cohorts.
  Route of administration: Oral Dose interval and frequency: Once daily for 7 days
  Arms: Part 2 MAD
Drug: Placebo — Matching placebo will be administered across SAD and MAD
  Arms: Placebo

SUMMARY:
This is a first-in-human (FIH) study to evaluate the safety, tolerability, and pharmacokinetics (PK) of single and multiple ascending oral doses of HC002 in healthy adult participants.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, placebo-controlled, two-part study to evaluate the safety, tolerability, and PK of single (Part 1) and multiple (Part 2) oral doses of HC002.

The study will enroll approximately 56 participants across 2 parts. In Part 1 (SAD), there will be 4 cohorts and in Part 2 (MAD), there will be 3 cohorts. In Part 1, a single dose of HC002 or placebo will be administered on Day 1. In Part 2, multiple doses of HC002 or placebo will be administered once daily (QD) from Day 1 to Day 7.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants of 18 to 65 years of age (inclusive)
2. Able to read, understand, sign, and date a written informed consent form (ICF) before study participation at Screening
3. Male participants must agree to use accepted contraceptive regimens during the study and for a period after the last drug administration.
4. Female participants must not be pregnant, intending to become pregnant, or be lactating at any time during the study, and must agree to use accepted contraceptive regimens during the study and for a period after the last drug administration.
5. Body mass index (BMI) between 18.0 and 35.0 kg/m2 (inclusive) at screening and body weight ≥ 50 kg.
6. Judged to be in good health on the basis of medical history, physical examination, and routine laboratory measurements (i.e., without clinically relevant pathology).
7. No clinically significant findings on electrocardiogram (ECG) (12-lead), arterial blood pressure, or heart rate as determined at the discretion of the Investigator.
8. Non-smoker, ex-smoker (being defined as persons who completely stopped smoking cigarettes for at least 6 months), or social smoker (being defined as persons who smoke fewer than the equivalent of 10 nicotine containing products per month).
9. Able to understand and comply with protocol requirements and instructions and likely to complete the study as planned at Screening and upon admission as per PI's judgement.

Exclusion Criteria:

1. History of any illness or condition that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant.
2. Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with PK of the study drug (except appendectomy, hemorrhoidectomy and simple hernia repair).
3. Regular treatment with prescription or nonprescription medications which, at the discretion of the Investigator, may impact either participant safety during the trial or the study objectives. The continued use of prescribed hormonal contraceptives is permitted, provided use has been stable for 3 months.
4. Consumption of herbal medications, dietary supplements, and specific fruit products (ie, pomello, Seville orange, and grapefruit).
5. History of drug addiction within 2 years before the start of study drug dosing, or a positive test result for drugs of abuse, such as tetrahydrocannabinol (THC), cocaine, amphetamines, barbiturates, benzodiazepines, opiates, methadone, methamphetamines, methylenedioxymethamphetamine (MDMA), and phencyclidine (PCP).
6. History of alcohol addiction within 2 years before the start of study drug dosing, positive test for alcohol, or engages in regular consumption of more than 4 units of alcoholic beverages per day or more than 10 units per week (1 unit of alcohol is equivalent to approximately 1 pint [473 mL] of beer or lager, 1 glass [125 mL] of wine, or 25 mL shot of 40% spirit) before Screening.
7. Participation in a clinical study involving administration of either an investigational or a marketed drug within 30 days, 5 half-lives, or until the expected pharmacodynamic effect has returned to Baseline (whichever is longer) before Screening.
8. Blood donation or a significant loss of blood within 60 days of the start of study drug dosing or donation of more than 1 unit of plasma within 7 days before Screening.
9. Positive result at Screening for any of the following infectious disease tests: hepatitis A virus, hepatitis B virus, hepatitis C virus, and human immunodeficiency virus (HIV-1/-2).
10. Illness within 5 days before the start of study drug dosing ("illness" is defined as an acute [serious or non-serious] condition [e.g., the flu or the common cold]).
11. History of any known relevant allergy/hypersensitivity (including allergy to the study drug or its excipients).
12. Suicidal tendency, history of or disposition to seizures, state of confusion, and/or a diagnosis with a clinically relevant psychiatric disease.
13. Use of immunotherapy within 3 months prior to Screening.
14. Abnormal liver function (ALT > 1.5-times upper limit of normal (ULN) or bilirubin > 1.5-times ULN).
15. Prescence of out-of-range cardiac interval (HR 45 to 100 beats per minute, PR 120 to 220 msec, QRS < 120 msec, and QTcB ≤ 470 msec [female] or ≤ 450 msec [male]) on the Screening ECG or other clinically significant ECG abnormalities as determined by the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
To assess the safety of HC002 by the incidence of adverse events | SAD- Screening to Day 4 post first dose administration; MAD- screening to Day 11 post first dose administration
Number of participants with abnormal laboratory values and/or adverse events that are related to treatment | SAD- Screening to Day 4 post first dose administration; MAD- screening to Day 11 post first dose administration
Number of participants with changes to the electrocardiogram (ECG) from baseline recorded as adverse events | SAD- Screening to Day 4 post first dose administration; MAD- screening to Day 11 post first dose administration

SECONDARY OUTCOMES:
Plasma PK parameters- Maximum plasma concentration (Cmax) after first dose of HC002 | SAD-Samples will be collected on Day 1 to Day 3 post first dose administration; MAD-Samples collected across 11 timepoints on Day 1 and Day 7 post first dose administration
Plasma PK parameters- Time for maximum plasma concentration (Tmax) after first dose of HC002 | SAD-Samples will be collected on Day 1 to Day 3 post first dose administration; MAD-Samples collected across 11 timepoints on Day 1 and Day 7 post first dose administration
Plasma PK parameters-- Area under curve (AUC) after first dose of HC002 | SAD-Samples will be collected on Day 1 to Day 3 post first dose administration; MAD-Samples collected across 11 timepoints on Day 1 and Day 7 post first dose administration
Plasma PK parameters- Apparent clearance (CL/F) after first dose of HC002 | SAD-Samples will be collected on Day 1 to Day 3 post first dose administration; MAD-Samples collected across 11 timepoints on Day 1 and Day 7 post first dose administration
Plasma PK parameters- terminal half-life (t1/2) after first dose of HC002 | SAD-Samples will be collected on Day 1 to Day 3 post first dose administration; MAD-Samples collected across 11 timepoints on Day 1 and Day 7 post first dose administration
Plasma PK parameters- Vz/F (apparent volume of distribution) after first dose of HC002 | SAD-Samples will be collected on Day 1 to Day 3 post first dose administration; MAD-Samples collected across 11 timepoints on Day 1 and Day 7 post first dose administration
Urine PK parameters- Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) after first dose of HC002 | SAD-Samples will be collected 4 timepoints from Day1 to Day 2 post first dose administration; MAD- Samples collected across 5 time-intervals from Day 1 to Day 7 post first dose administration]
Urine PK parameters- fet1-t2 (fraction of analyte excreted in urine from time point t1 to t2) after first dose of HC002 | SAD-Samples will be collected 4 timepoints from Day1 to Day 2 post first dose administration; MAD- Samples collected across 5 time-intervals from Day 1 to Day 7 post first dose administration
Urine PK parameters-Clearance rate (CLr) after first dose of HC002 | SAD-Samples will be collected 4 timepoints from Day1 to Day 2 post first dose administration; MAD- Samples collected across 5 time-intervals from Day 1 to Day 7 post first dose administration

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No